CLINICAL TRIAL: NCT04613037
Title: Efficacy of Fecal Microbial Transplantation Treatment in Adults With Atopic Dermatitis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0452-17
Record Dates: First submitted 2020-10-15; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Prospective single-blinded placebo-controlled cross-over study, among adult patients suffering from moderate-to-severe atopic dermatitis (AD), insufficiently responsive to topical and systemic treatment. All patients receive 2 placebo transplantations each 2 weeks apart followed by 4 fecal microbial transplantations (FMTs) from healthy donors each 2 weeks apart. Patients were allowed to continue with their baseline medical topical treatment, including moisturizers and glucocorticoids, during the study period, but no new therapy was commenced
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Fecal Microbial Transplantation in adults with Atopic Dermatitis
  Interventions: Biological: Fecal Microbial Transplantation

INTERVENTIONS:
Biological: Fecal Microbial Transplantation — Fecal Microbial Transplantation in adults with Atopic Dermatitis

SUMMARY:
Prospective single-blinded placebo-controlled cross-over study, among adult patients suffering from moderate-to-severe atopic dermatitis (AD), insufficiently responsive to topical and systemic treatment. All patients receive 2 placebo transplantations each 2 weeks apart followed by 4 fecal microbial transplantations (FMTs) from healthy donors each 2 weeks apart. Patients were allowed to continue with their baseline medical topical treatment, including moisturizers and glucocorticoids, during the study period, but no new therapy was commenced. The severity of AD and the fecal microbiome profile was evaluated by the Scoring Atopic Dermatitis Score (SCORAD score), and the weekly use of topical corticosteroids, at the beginning of the study, before every FMT, and 1-6 months after the last FMT.

DETAILED DESCRIPTION:
Prospective single-blinded placebo-controlled cross-over study, among adult patients suffering from moderate-to-severe atopic dermatitis (AD), insufficiently responsive to topical and systemic treatment. All patients receive 2 placebo transplantations each 2 weeks apart followed by 4 fecal microbial transplantations (FMTs) from healthy donors each 2 weeks apart. Patients were allowed to continue with their baseline medical topical treatment, including moisturizers and glucocorticoids, during the study period, but no new therapy was commenced. The severity of AD and the fecal microbiome profile were evaluated by the Scoring Atopic Dermatitis Score (SCORAD score), and the weekly use of topical corticosteroids, at the beginning of the study, before every FMT, and 1-6 months after the last FMT.

During the study period, patients were allowed to use only topical therapy including emollients and glucocorticoids or calcineurin inhibitors.

FMT preparation and delivery:

Volunteer donors were healthy, non-pregnant adults aged 18 to 50 years, with a normal body mass index. Volunteer donors were excluded for any significant medical history or for any use of antibiotics in the preceding 3 months. Candidates were eligible according to the Israeli Ministry of Health guidelines which include a physical examination and laboratory screening tests including fecal enteric pathogens, serum antibodies to hepatitis A, B, and C; human immunodeficiency virus; HTLV, and Treponema pallidum as well as celiac, CBC (and additional tests that comply with the guidelines of the Israeli Ministry of Health). Stool was delivered within minutes post defecation in a clean closed plastic container and was processed at the Tel Aviv Medical Center stool bank facility to prepare capsulized FMT. Briefly, fecal material was diluted with normal saline (600ml/100g of fecal material), filtered and concentrated the preparation in a centrifuge. The pellet was suspended in sterile saline and glycerol (20%) that was added as a bacterial cryoprotectant. This material was then pipetted into acid-resistant capsules, which was closed and then secondarily sealed with additional set of capsules. Capsules were stored frozen at -80°C. Placebo capsules had identical visually and contained diluted glycerol only.

Capsulized FMT procedure:

FMT was administered in two doses of 15 FMT capsules on two consecutive days (a total of 30 capsules), at the Bacteriotherapy clinic of the Tel Aviv medical center (TLVMC). On the day of administration, capsules frozen at -80°C were taken out of the freezer and transported to the clinic on ice. Fifteen capsules were handed individually to the patient and the patient ingested the capsules immediately with some water. Patients were asked to fast overnight prior to capsule intake.

Fecal microbial analysis:

In order to examine whether the clinical effect may be mediated by colonization of new bacterial strains, the investigators developed a robust and sensitive method to calculate pairwise DNA sequence dissimilarity between bacterial strains of the same species across distinct metagenomics samples. Donor stool samples that were used for FMT capsules and stool samples that were collected from the patients during the study period were sequenced into metagenomics reads. Reads that were mapped were piled up to obtain per-position variant information for every detected species. Difference in the variant of a particular species at a given position between two samples was defined as having no intersection between the set of detected alleles in the two samples being compared. The estimated species DNA sequence dissimilarity for a pair of samples is then the number of different positions divided by the total number of positions being compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are ≥18 years of age
* Moderate-to-severe atopic dermatitis, as defined by a Scoring Atopic Dermatitis Score (SCORAD) score ≥25
* Disease duration minimum of 3 years that was inadequately controlled by topical and systemic therapy

Exclusion Criteria:

* Age under 18 years
* Pregnancy
* Another concomitant active dermatologic disease.
* Receiving systemic therapy including phototherapy within 4 weeks before the beginning of the study.
* Receiving any antibiotic or probiotic treatment within 4 weeks before the beginning of the study or during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Assessment of the change in the severity of Atopic Dermatitis after treatment with Fecal Microbial Transplantation | 2 weeks after each FMT, and 8 weeks or more after the last FMT
  Overall mean change from baseline of the Scoring atopic dermatitis score (SCORAD), described and validated by the European Task Force on Atopic Dermatitis, used for the assessment of the severity of Atopic Dermatitis. The minimal SCORAD score, describing a situation without any signs of atopic dermatitis is 0, the disease is not visible, while the maximal score, describing the most severe presentation of atopic dermatitis, is 103.

SECONDARY OUTCOMES:
Assessment of the degree of bacterial strain transmission from donor to patient after treatment with Fecal Microbial Transplantation | 2 weeks after each FMT, and 8 weeks or more after the last FMT
  Fecal microbial species in donors' and in patients' stool were assessed after each FMT. A metagenomics analysis (Illumina NextSeq) was used to assess the microbial strain distribution in each fecal sample. Patient-donor dissimilarities across different study time points were compared to intra-host dissimilarities in a healthy reference population. Transmission was defined as a dissimilarity between two strains among donor and recipient above the detection threshold of 5e-5.
Assessment of the correlation between bacterial stains transmission from donor to patient to the SCORAD score change after treatment with Fecal Microbial Transplantation | 2 weeks after each FMT, and 8 weeks or more after the last FMT
  The change in disease severity (SCORAD score change) was correlated with samples strains dissimilarities between donors and their recipients (Pearson correlation method) to evaluate whether there was a correlation between the degree of strain transmission to the clinical improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Mashiah, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center; Nitsan Maharshak, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Department of Dermatology, Tel Aviv Sourasky medical center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Yes
After termination of the study protocol for all participants the data and stool and blood samples was shared in order to perform fecal microbial analysis to examine whether the clinical effect may be mediated by colonization of new bacterial strains
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After termination of the study protocol for all participants the data and stool and blood samples were shared
Access Criteria: All information was given to the researcher that performed the fecal microbial analysis